CLINICAL TRIAL: NCT05260034
Title: Minimizing Fall-Related Injury in Older Adults: a Motor Learning Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00147362; R21AG073892 (NIH)
Record Dates: First submitted 2022-01-24; First posted 2022-03-02 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Fall Injury; Fall Patients; Mobility Limitation
Keywords: Falls; Physical Therapy; Injury Prevention
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: In the current study, participants and intervention trainers are unmasked to the treatment and know which group they are working on. Only the assessor will be masked to the groups of participants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Otago Group (Active Comparator): The control group will receive balance exercises adapted from the evidenced-based Otago Exercise program. Briefly, all eight sessions (~30 min) will involve balance exercises and strength exercises using ankle weights, and will progressively increase as performance improves by increasing resistance or the difficulty of the balance exercises (e.g., reducing base of support).
  Interventions: Other: Otago Exercise Program
- FAST Group (Experimental): Participants randomized to the intervention arm will undergo the FAST program, a progressive safe-falling training based on the tuck and roll strategy. As part of the FAST program, participants will train 30 minutes twice a week for a period of four weeks under the supervision of a trained researcher. Participants will wear protective gear (knee, hip, head) and they will complete a 10-minute stretching exercise routine to minimize the risk of injury.
  Interventions: Other: FAST Program

INTERVENTIONS:
Other: FAST Program — This program aims to teach how to effectively reduce impact forces during a sideways fall by 1) changing the trunk/knee angles during descent to decrease body acceleration, 2) using a rolling movement to allow for an optimal distribution of impact forces applied to any site along the contact path; and 3) tucking the chin to protect the head.
  Arms: FAST Group
Other: Otago Exercise Program — The Otago Exercise Program (OEP) was chosen, rather than no control intervention, to increase the level of evidence required to demonstrate efficacy, and because, similar to the safe fall training used here, it was designed to be performed individually or in small groups.
  Arms: Otago Group

SUMMARY:
Falls are the leading cause of accidental injury and injury-related death among older adults. Despite evidence that falls can be prevented, fall related injuries have not declined over time. Current fall injury prevention techniques targeting mobility and bone strength have merit yet their effectiveness is limited. Indeed, a recent Patient Centered Outcomes Research Institute/National Institute on Aging funded pragmatic trial of individualized multifactorial strategy to prevent serious fall injuries in over 5500 seniors revealed no difference in fall injuries between the intervention and standard care arm. The inconclusive results of the investigation may be due in part to focusing on fall prevention rather than mitigation of fall-related impact acceleration and forces - the "fundamental variables" for injury prevention. A fall-related injury occurs when the body hits the ground with force that is greater than tissue strength. Development of innovative approaches that focus on fundamental variables of injury prevention is needed.

DETAILED DESCRIPTION:
Impact forces and body accelerations can be mitigated by performing specific movement patterns during the impact phase of a fall. The investigators, along with others have postulated and provided preliminary evidence that older adults can learn specific movement patterns (enacted during the impact phase of a fall), such as the tuck and roll that significantly reduce impact forces and minimize the risk of injury. The investigators' recent Randomized Clinical Trial (RCT) that examined the FAlling Safely Training (FAST) program in 17 older adults with low fall risk found that following 2 hours of training, the FAST group reduced their hip impact force by 33% and head acceleration by 59% and demonstrated retention. The procedures were feasible and safe in relatively healthy older adults with low fall risk. Despite the promise of this approach, perhaps the most important issue for real world translation is whether at-fall risk older adults with known balance impairment, a key target group who would most benefit from this training, can safely learn to fall with reduced impact forces and thus potentially fewer injuries using this paradigm. The immediate goal of this investigation is to determine the safety and feasibility of FAST training in an at-fall risk older adult group, the key measurable stages of FAST mastery, and, most importantly, the effect size, compared to modified Otago Exercise Program (an evidence-based fall risk reduction program) controls, to inform a larger future trial. To maximize safety, participants will utilize a protective helmet, and hip protector while landing on a cushioned pad. In addition, using a motor learning approach, the investigators will determine and measure key stages of the technique that can be mastered and measured as intermediate measures to document training progression.

ELIGIBILITY:
Inclusion Criteria:

* Have balance impairment as indicated by <10s on unipedal stance
* History of fall injury in the last year; or, two more falls in the last year; or, afraid of falling because of problems with balance or walking
* Have no history of tumbling, gymnastic or martial art experience or currently engagement of 150+ minutes/week of vigorour aerobic activity
* No clinical osteoporosis
* DEXA (dual energy X-ray absorptiometry) determined bone mineral density of the hip of t is greater than or equal to -2.3

Exclusion Criteria:

* Outside of age range
* Unable to speak or comprehend written/spoken English
* Cognitive impairment as indicated by Saint Louis University Memory Scale (<25)
* Unable to ambulate household distances
* Intact standing balance as indicated by >10s of unipedal stance
* Currently receiving physical therapy
* Presence of clinical osteoporosis
* Uncorrected vision or hearing or vestibular dysfunction
* Major neurological conditions, such as stroke, Parkinson's Disease, vertigo that affect the ability to ambulate or perform daily tasks
* Currently taking medications, including, coumadin, dual oral anticoagulants (apixaban, rivaroxaban), lovenox
* Conditions may lead to (internal) bleeding, such as thrombocytopenia, hemorrhagic diathesis

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
Physical discomfort related to the intervention | The physical discomfort scale will be utilized through the participant's involvement in the study, approximately five months.
  The hypothesis is that there will be minimally greater musculoskeletal discomfort in the FAST group that than in the Otago Exercise Program group, but no difference in adverse events. Physical discomfort will be recorded by an 11-point numerical rating scale (ranging from 0, no discomfort to 10, worst imaginable discomfort). Participants will self-report their discomfort, including the physical location and severity on a standardized body map.
Participant ability to master the intervention | Feasibility will be measured during the intervention, which will last four weeks.
  The investigators hypothesize that at least 2/3 of FAST participants will pass through a series of technique mastery and eventually progress to the final stage of the training. Mastery of technique will be measured by scoring the participants' technique based on predetermined, standardized competency criteria.
Determining FAST efficacy in reducing hip impact force, versus Otago Exercise Program (OEP). | The outcome will measured at the baseline, one-week post-intervention, and three-months post-intervention.
  The first part of the hypothesis postulates that when compared to baseline, FAST participants will show greater reduction in hip impact force than OEP participants immediately post-training. The second part of the hypothesis postulates that compared to baseline, FAST participants will show greater reduction in hip impact force than OEP participants at three months post-training. The impact velocity and impact acceleration of the hip will be computed based on the hip trajectory recorded by motion capture system.
Determining FAST efficacy in reducing head acceleration, versus Otago Exercise Program (OEP). | The outcome will be measured during the baseline, one-week post-intervention, and three-months post-intervention.
  The first part of the hypothesis postulates that when compared to baseline, FAST participants will show greater reduction in head acceleration than OEP participants immediately post-training. The second part of the hypothesis postulates that compared to baseline, FAST participants will show greater reduction in head acceleration than OEP participants at three months post-training. Information will be collected on upper limb impact by utilizing conformal sensors during falls.
Number of adverse events | AEs and SAEs will be monitored through participant involvement of the study, approximately five months.
  Any adverse events (AEs) and serious adverse events (SAEs) will be recorded on the Council for International Organizations of Medical Sciences' CIOMS-E2A form by the researchers. The definition of adverse event and serious adverse events will follow that of the International Council for Harmonization.

SECONDARY OUTCOMES:
The number of head impacts | The outcome will be measured during the baseline, one-week post-intervention, and three-months post-intervention.
  The number of times that the head makes contact with the ground will be recorded at each assessment.
The movement strategy of falls | The trunk angle, knee angle and trunk rotation of each fall will be assessed at all assessments (baseline, one-week post-intervention, and 3-month follow-up).
  The trunk angle, knee angle and trunk rotation at impact will be calculated based on the motion capture data, which will measure the body's angles and rotation during the fall. Each assessment will have the right and left side falls for 2 trials each and 2 backward falls, in a total.

OTHER OUTCOMES:
Balance | BBS will be assessed at all assessments (baseline, one-week post-intervention, and 3-month follow-up). Each assessment will last about 1.5 hours.
  Balance will be quantified by the Berg Balance Scale (BBS). This is a 14-item object measure of static balance and fall risk in older adults. The 14 items range from quiet standing, to sit to stand, to tandem standing. Each item is scored 0-4 (unable to complete to successful completion) and the item scores are summed with a total of 56 for maximal performance.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Sosnoff, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- Emma Eells, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zanotto A, Zanotto T, Alexander NB, Sosnoff JJ. Views and experiences of older people taking part in a safe-falling training program: Lessons learned from the FAlling Safely Training (FAST) trial. BMC Geriatr. 2024 Oct 11;24(1):818. doi: 10.1186/s12877-024-05382-7. PMID 39394576
- [Derived] Zanotto T, Chen L, Fang J, Bhattacharya SB, Alexander NB, Sosnoff JJ. Minimizing fall-related injuries in at-risk older adults: The falling safely training (FAST) study protocol. Contemp Clin Trials Commun. 2023 Apr 11;33:101133. doi: 10.1016/j.conctc.2023.101133. eCollection 2023 Jun. PMID 37122489